CLINICAL TRIAL: NCT02526745
Title: Safety and Immunogenicity Study of Live Attenuated Vaccine Against Herpes Zoster in Chinese Adults Aged 50 Years and Older
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Chaoyang District Centre for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: cycdc2015-1
Record Dates: First submitted 2015-08-12; First posted 2015-08-18 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2015-08

CONDITIONS: Herpes Zoster
Keywords: vaccine; safety; immunogenicity
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- high doses of virus content between 4.7～5.0 lgPFU (Experimental): live attenuated vaccine against herpes zoster with high doses of virus content between 4.7～5.0 lgPFU in 20 adults aged 50-80 years old on day 0
  Interventions: Biological: the vaccine with high doses of virus content between 4.7～5.0 lgPFU
- low doses of virus content between 4.7～5.0 lgPFU (Experimental): live attenuated vaccine against herpes zoster with low doses of virus content between 4.7～5.0 lgPFU in 20 adults aged 50-80 years old on day 0
  Interventions: Biological: the vaccine with low doses of virus content between 4.7～5.0 lgPFU
- high doses of virus content between 4.3～5.0 lgPFU (Experimental): live attenuated vaccine against herpes zoster with high doses of virus content between 4.3～5.0 lgPFU in 100 adults aged 50-80 years old on day 0
  Interventions: Biological: the vaccine with high doses of virus content between 4.3～5.0 lgPFU
- middle doses of virus content between 4.3～5.0 lgPFU (Experimental): live attenuated vaccine against herpes zoster with middle doses of virus content between 4.3～5.0 lgPFU in 100 adults aged 50-80 years old on day 0
  Interventions: Biological: the vaccine with middle doses of virus content between 4.3～5.0 lgPFU
- low doses of virus content between 4.3～5.0 lgPFU (Experimental): live attenuated vaccine against herpes zoster with low doses of virus content between 4.3～5.0 lgPFU in 100 adults aged 50-80 years old on day 0
  Interventions: Biological: the vaccine with low doses of virus content between 4.3～5.0 lgPFU
- placebo (Placebo Comparator): placebo in 100 adults aged 50-80 years old on day 0
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: the vaccine with high doses of virus content between 4.7～5.0 lgPFU
  Arms: high doses of virus content between 4.7～5.0 lgPFU
Biological: the vaccine with low doses of virus content between 4.7～5.0 lgPFU
  Arms: low doses of virus content between 4.7～5.0 lgPFU
Biological: the vaccine with high doses of virus content between 4.3～5.0 lgPFU
  Arms: high doses of virus content between 4.3～5.0 lgPFU
Biological: the vaccine with middle doses of virus content between 4.3～5.0 lgPFU
  Arms: middle doses of virus content between 4.3～5.0 lgPFU
Biological: the vaccine with low doses of virus content between 4.3～5.0 lgPFU
  Arms: low doses of virus content between 4.3～5.0 lgPFU
Biological: placebo
  Arms: placebo

SUMMARY:
This study evaluates the safety and immunogenicity of live attenuated vaccine in adults aged 50 years and older. Half of participants will receive high doses of the vaccine,while the other half will receive low doses of the vaccine in phase I clinical trial. At the phase II clinical trial, participants will be distributed equally to four groups(low、middle, high doses of the vaccine and placebo).

ELIGIBILITY:
Inclusion Criteria:

* Adults 50 years and older,no vaccine contraindications;
* Subject to comply with the requirements of clinical trial programs;
* No immune globulin vaccination history within a month, no vaccination history within 28 days;
* Axillary temperature ≤37.0 ℃;
* Patients with chronic diseases should be in stable ;
* Postmenopausal or female subjects is no longer the possibility of pregnancy, or subjects pregnancy test was negative and has no pregnancy planner during the clinical trial period;
* The value of blood routine (WBC, RBC, Hb) is normal , or abnormal but meaningless by clinicians judgment ;
* Alanine aminotransferase (ALT) values is normal, or abnormal but meaningless by clinicians judgment ;
* Renal function (serum urea nitrogen) is normal, or abnormal but meaningless by clinicians judgment.

Exclusion Criteria:

* Allergies, seizures, epilepsy, encephalopathy and other medical history or family history of mental illness;
* Subjects who is allergic to any element of the vaccine,and have a history of severe allergy to any vaccine;
* Subjects who is suffering from immune deficiency, receiving immunosuppressive therapy or immunocompromised due to HIV;
* Subjects who had a history of herpes zoster five years ago;
* Varicella or herpes zoster vaccination history;
* Pregnant or lactating women;
* Women who are planning a pregnancy in the near future;
* Any prior administration of vaccine in last 28 days or planned to vaccinate any vaccine during the observation period;
* Suffering from acute febrile diseases, and infectious diseases;
* Thrombocytopenia or other coagulation disorder history, which may cause subcutaneous taboo;
* Accept any other investigational drug users within two months;
* Subjects had high fever (axillary temperature ≥38.0 ℃) in the past three days ;
* The value of blood routine (WBC, RBC, Hb) is abnormal and meaning by clinicians judgment ;
* Alanine aminotransferase (ALT) values is abnormal and meaning by clinicians judgment ;
* Renal function (serum urea nitrogen) is abnormal and meaning by clinicians judgment.
* Blood pressure is abnormal after medication control;
* Known or suspected diseases including: respiratory diseases, acute infection or chronic disease , and cardiovascular disease, kidney disease, skin disorders in the acute phase;
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2015-12; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the Rate of Adverse reactions of live attenuated Herpes zoster Vaccine in Chinese Adults. | 42 days
  Adverse reactions associated with vaccine will be observed in Chinese Adults ( 50 years and older) after vaccination. Solicited local adverse events include Pain, Redness, Swelling, Induration, Rash, Pruritus at injection site. solicited general adverse events include Fever, Nausea, Vomiting, Diarrhea, Decreased appetite, Be agitated (irritability, abnormal crying), fatigue, allergy

SECONDARY OUTCOMES:
Evaluate the seroconversion rate of anti-herpes zoster virus antibodies in serum of adults after vaccination. | 6 months
  The seroconversion rate of anti-herpes zoster virus antibodies will be evaluated in serum of adults within the first 42 days after vaccination.

REFERENCES:
- [Derived] de Oliveira Gomes J, Gagliardi AM, Andriolo BN, Torloni MR, Andriolo RB, Puga MEDS, Canteiro Cruz E. Vaccines for preventing herpes zoster in older adults. Cochrane Database Syst Rev. 2023 Oct 2;10(10):CD008858. doi: 10.1002/14651858.CD008858.pub5. PMID 37781954